CLINICAL TRIAL: NCT04601805
Title: Optical Coherence Tomography Angiography Assessment of Retinal Lesions in Inflammatory Bowel Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Dina Tadros, Lecturer of Ophthalmology, Tanta University, Egypt, Tanta University
Other Study IDs: 34002/8/20
Record Dates: First submitted 2020-10-13; First posted 2020-10-26 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Group (1) : Patient diagnosed with IBD with no treatment received
  Interventions: Device: Observation
- Group(2): Patient diagnosed with IBD and received treatment for a long time
  Interventions: Device: Observation

INTERVENTIONS:
Device: Observation — We will record the vascular changes that follow the inflammatory bowel diseases

SUMMARY:
Aim of the study;To record the vascular changes that may be present in the posterior segment of patients suffering from Inflammatory bowel diseases(IBD) using the optical coherence tomography angiography

DETAILED DESCRIPTION:
a prospective study of 30 patients suffering from IBD referred from tropical department from Tanta University Hospital

-Patients demographic data e.g., sex, age, concomitant systemic diseases will be recruited. Presenting symptoms, physical examination results, laboratory and imaging findings, and received treatment of IBD will be recorded. Accurate grading of disease severity will be carried out by gastroenterology specialist.

All patients will be subject to Full ophthalmologic examination and fundus imaging. Imaging will include OCTA and fundus photography. OCTA will be performed using cirrus OCT (Zeiss, Inc., USA). High-quality 6 x 6 mm OCTA macular scans and 3 × 3-mm papillary scan with strong signal-noise ratio and adequate centration on the fovea and optic nerve head respectively will be selected. Segmentation will be used to evaluate superﬁcial and deep capillary retinal plexus projections in addition to the choriocapillaries. If errors in segmentation were detected, manual correction would be performed. The superﬁcial retinal capillary plexus (SCP) will be delineated with an inner boundary at the internal limiting membrane (ILM) and an outer boundary 10 µm inside the inner plexiform layer (IPL). The deep retinal capillary plexus (DCP) will be segmented with an inner boundary 10 µm inside the IPL and an outer boundary at 10 µm beneath the outer plexiform layer (OPL).

The vessel density metric from enface OCT angiogram will be used as an indicator of macular retinal and papillary perfusion. Vessel density (VD) analysis computes the percentage of area occupied by OCTA detected vasculature in a measured area. Choriocapillaries flow voids will be computed to assess choriocapillaries circulation

ELIGIBILITY:
Inclusion Criteria:

* Patients with Crohn's disease and ulcerative colitis either newly diagnosed or suffering from chronic disease on treatment will be included

Exclusion Criteria:

* Recent ophthalmological surgery.

  * Low quality ophthalmological exams.
  * Refractive errors greater than + 3 or - 3 spherical.
  * Retinopathies such as diabetic retinopathy.
  * Any type of retinal degenerations or retinal dystrophy.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This will be a prospective study of 30 patients suffering from Inflammatory bowel disease referred from tropical department from Tanta University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-04-13 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2024-12-29 (Estimated)

PRIMARY OUTCOMES:
vascular changes in the posterior segment of patients suffering from inflammatory bowel disease using the optical coherence tomography angiography | 1 month
  OCTA will be performed using cirrus OCT (Zeiss, Inc., USA). High-quality 6 x 6 mm OCTA macular scans and 3 × 3-mm papillary scan with strong signal-noise ratio withadequate centration on the fovea and optic nerve head Segmentation will be used to evaluate superﬁcial and deep capillary retinal plexus projections in addition to the choriocapillaries. The superﬁcial retinal capillary plexus (SCP) will be delineated with an inner boundary at the internal limiting membrane (ILM) and an outer boundary 10 µm inside the inner plexiform layer (IPL). The deep retinal capillary plexus (DCP) will be segmented with an inner boundary 10 µm inside the IPL and an outer boundary at 10 µm beneath the outer plexiform layer (OPL).
  The vessel density metric from enface OCT angiogram as an indicator of macular retinal and papillary perfusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospital, Tanta, El-Garbeia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Silva FA, Rodrigues BL, Ayrizono ML, Leal RF. The Immunological Basis of Inflammatory Bowel Disease. Gastroenterol Res Pract. 2016;2016:2097274. doi: 10.1155/2016/2097274. Epub 2016 Dec 14. PMID 28070181
- [Result] Zhang YZ, Li YY. Inflammatory bowel disease: pathogenesis. World J Gastroenterol. 2014 Jan 7;20(1):91-9. doi: 10.3748/wjg.v20.i1.91. PMID 24415861
- [Result] Ghanchi FD, Rembacken BJ. Inflammatory bowel disease and the eye. Surv Ophthalmol. 2003 Nov-Dec;48(6):663-76. doi: 10.1016/j.survophthal.2003.08.004. PMID 14609712
- [Result] Troncoso LL, Biancardi AL, de Moraes HV Jr, Zaltman C. Ophthalmic manifestations in patients with inflammatory bowel disease: A review. World J Gastroenterol. 2017 Aug 28;23(32):5836-5848. doi: 10.3748/wjg.v23.i32.5836. PMID 28932076
- [Result] Familiari L, Strangio G, Consolo P, Luigiano C, Bonica M, Barresi G, Barresi V, Familiari P, D'Arrigo G, Alibrandi A, Zirilli A, Fries W, Scaffidi M. Optical coherence tomography evaluation of ulcerative colitis: the patterns and the comparison with histology. Am J Gastroenterol. 2006 Dec;101(12):2833-40. doi: 10.1111/j.1572-0241.2006.00826.x. PMID 17227526
- [Result] Yilmaz S, Aydemir E, Maden A, Unsal B. The prevalence of ocular involvement in patients with inflammatory bowel disease. Int J Colorectal Dis. 2007 Sep;22(9):1027-30. doi: 10.1007/s00384-007-0275-1. Epub 2007 Jan 30. PMID 17262200
- [Result] Or C, Sabrosa AS, Sorour O, Arya M, Waheed N. Use of OCTA, FA, and Ultra-Widefield Imaging in Quantifying Retinal Ischemia: A Review. Asia Pac J Ophthalmol (Phila). 2018 Jan-Feb;7(1):46-51. doi: 10.22608/APO.201812. Epub 2018 Feb 13. PMID 29436208